CLINICAL TRIAL: NCT01134692
Title: COMPARATIVE STUDY OF NORFLOXACIN AND PROBIOTICS ON PORTAL PRESSURE IN PATIENTS WITH CIRRHOSIS AND LARGE VARICES WHO HAVE NEVER BLED IN THE PAST
Brief Title: Probiotics for Portal Hypertension
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Govind Ballabh Pant Hospital (Other Government)
Responsible Party: Nitin Gupta, G.B. Pant Hospital, Delhi
Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NG002
Record Dates: First submitted 2010-06-01; First posted 2010-06-02 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-05

CONDITIONS: Cirrhosis; Varices, Esophageal
Keywords: Patients with cirrhosis who have large esophageal varices with No history of upper GI bleeding in the past
MeSH Terms: conditions — Fibrosis; Esophageal and Gastric Varices | interventions — Propranolol; Norfloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Propranolol + Placebo (Placebo Comparator)
  Interventions: Drug: Propranolol, Norfloxacin, VSL#3
- Propranolol + Norfloxacin (Active Comparator): drug
  Interventions: Drug: Propranolol, Norfloxacin, VSL#3
- Propranolol + Probiotic (Experimental): VSL#3
  Interventions: Drug: Propranolol, Norfloxacin, VSL#3

INTERVENTIONS:
Drug: Propranolol, Norfloxacin, VSL#3 — Propranolol: as per heart rate titration Norfloxacin: 400mg BD

SUMMARY:
Chronic peripheral and splanchnic vasodilatation are the hallmark hemodynamic abnormality in cirrhosis and contribute to the pathogenesis of portal hypertension.

Alterations in intestinal motility and bacterial overgrowth in gut may predispose to the development of bacteraemia and endotoxaemia in cirrhotic patients which play a role in the hyperdynamic circulatory syndrome of cirrhosis. Probiotic therapy is aimed at changing the make-up of the indigenous microflora by administering specific strains of non-pathogenic and potentially beneficial microflora. In this study, the investigators hypothesize that a modification in the composition of the endogenous digestive microflora by oral bacteriotherapy with high potency probiotic preparations could be a safe way to regulate the portal pressure.

As there is a relative paucity in effective pharmacological treatment for portal hypertension, these novel and innovative therapy might provide important alternative or adjunct therapy to beta blockers in the clinical management of patients with portal hypertension.

Aims and objectives

To study in patients with cirrhosis and large varices whether probiotics and/or norfloxacin given for 2 months :

1. achieve a reduction in HVPG
2. alter the endotoxin and cytokine levels, and improve systemic inflammatory responses
3. well tolerated.

Inclusion criteria:

Consecutive patients of cirrhosis with portal hypertension who fulfill the following criteria:

1. Diagnosed cases of cirrhosis (by clinical, biochemical and radiological criteria with or without liver biopsy)
2. No history of upper GI bleeding in the past
3. Endoscopically documented large esophageal varices

Exclusion criteria

1. history of gastrointestinal bleeding
2. patients who have received beta blockers for portal hypertension in the past 6 weeks.
3. hepatic encephalopathy
4. ongoing bacterial infection,
5. Spontaneous bacterial peritonitis
6. active alcoholism or illicit drug abuse
7. alcoholic hepatitis
8. Treatment with antibiotics in the preceding 2 weeks.
9. presence of hepatocellular carcinoma,
10. portal vein thrombosis
11. serum creatinine>1.5 mg/dL,
12. treatment with vasoactive drugs in the past 6 weeks,
13. history of arterial hypertension, congestive heart failure or arterial occlusive disease, and
14. Refusal to participate.
15. Active smokers.

Study plan:

Ethical approval will be obtained prior to study initiation. Patients presenting to Department of Gastroenterology, GB Pant Hospital will be recruited in the study. Patients will be evaluated regarding the eligibility for the study. After being found eligible for the study, if the patient agrees to participate in the study, a signed informed consent will be obtained. Baseline HVPG will be measured in all patients and then they will be randomized into 3 groups:.

1. Group 1: Beta blockers + placebo
2. Group 2: Beta blockers + Norfloxacin (400mg BD)
3. Group 3: Beta blockers + probiotics. (one sachet of VSL#3 BD)

30 patients will be enrolled into each group. The treatment will be continued for 2 months.

The study design is a randomized double-blinded placebo controlled trial.

Once patients have been enrolled, they will undergo baseline investigations. Blood will be drawn from both peripheral and hepatic veins and sent for routine parameters, pro-inflammatory cytokines (IL-1b, IL-6, IL-10, TNF-α, endotoxins, NO2 and NO3 levels, PRA, BNP). Samples will be stored at -70 ºC. Baseline vitals will be recorded.

Patients will be called at the end of 1 month for assessment of compliance and then at the end of the study (2 months) to repeat the HVPG and the same parameters as at the time of enrollment

End Points:

1. Primary

   a. Change in HVPG levels as compared with baseline, to define responder (≥20% reduction in HVPG or ≤ 12 mm Hg).
2. Secondary

   1. Change in digestive flora
   2. Reduction in serum and hepatic endotoxin and cytokine levels
   3. Assessment of improvement in the renal parameters and Systemic inflammatory response syndrome
   4. Improvement in the markers of oxidative injury
   5. Adverse effects

ELIGIBILITY:
Inclusion Criteria:

Consecutive patients of cirrhosis with portal hypertension who fulfill the following criteria:

1. Diagnosed cases of cirrhosis (by clinical, biochemical and radiological criteria with or without liver biopsy)
2. No history of upper GI bleeding in the past
3. Endoscopically documented large esophageal varices

Exclusion Criteria:

1. history of gastrointestinal bleeding
2. patients who have received beta blockers for portal hypertension in the past 6 weeks.
3. hepatic encephalopathy
4. ongoing bacterial infection,
5. Spontaneous bacterial peritonitis
6. active alcoholism or illicit drug abuse
7. alcoholic hepatitis
8. Treatment with antibiotics in the preceding 2 weeks.
9. presence of hepatocellular carcinoma,
10. portal vein thrombosis
11. serum creatinine>1.5 mg/dL,
12. treatment with vasoactive drugs in the past 6 weeks,
13. history of arterial hypertension, congestive heart failure or arterial occlusive disease, and
14. Refusal to participate.
15. Active smokers.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

PRIMARY OUTCOMES:
Change in HVPG levels as compared with baseline, to define responder (≥20% reduction in HVPG or ≤ 12 mm Hg). | 2 months

SECONDARY OUTCOMES:
Assessment of improvement in the renal parameters and Systemic inflammatory response syndrome | 2 months
Adverse effects | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- GB Pant hospital, Delhi, National Capital Territory of Delhi, India